CLINICAL TRIAL: NCT04551222
Title: Treatment of Veterans With Heart Failure With Reduced Ejection Fraction With Probenecid
Brief Title: The Re-Prosper HF Study
Acronym: Re-Prosper HF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARA-006-19F; I01CX001968 (NIH)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: heart failure; probenecid
MeSH Terms: conditions — Heart Failure | interventions — Probenecid

STUDY DESIGN:
Intervention Model Description: This is a three-site, double-blinded, randomized, placebo controlled, parallel design, trial in a 1:1 fashion of 1 gr. orally of probenecid twice daily or identical placebo for 180 days. The investigators propose to recruit 120 subjects (power analysis below) with HFrEF (LVEF 40%), NYHA II-III on guideline directed medical therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probenecid (Active Comparator): 1 gr. orally of probenecid twice daily for 180 days
  Interventions: Drug: probenecid
- Placebo (Placebo Comparator): identical placebo (to probenecid tablets) for 180 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: probenecid — 1 gr. orally of probenecid twice daily for 180 days
  Arms: Probenecid
Drug: Placebo — identical tablets to probenecid
  Arms: Placebo

SUMMARY:
Heart failure with reduced ejection fraction (HFrEF) is a common cause for admission within the Veterans Affairs (VA) Health Care System.

It is associated with severe impairment of physical and mental health status and carries a high risk of mortality. Even though significant progress has been made in understanding the disease process, currently, its management and treatment is limited.

The investigators have discovered that a commonly used drug for the treatment of gout can be repurposed for the treatment of HFrEF.

The objective of this study is the treatment of outpatient Veterans with HFrEF with probenecid to improve heart and health function. Specifically, the investigators are testing whether oral probenecid administered orally twice per day for 180 days improves heart function as measured via ultrasound of the heart (aim 1); improves exercise capacity (aim 2); and improves self-report heart failure specific health status as measured via questionnaires (aim 3).

DETAILED DESCRIPTION:
Heart failure with reduced ejection fraction (HFrEF) is a common cause for admission within the Veterans Affairs (VA) Health Care System. It is associated with severe impairment of physical and mental health status and carries a high 5-yr mortality rate of ~75%. Even though significant progress has been made in understanding its pathophysiology, currently, its management and treatment is based on therapeutic targeting of a limited number of receptors and pathways.

The investigators' team and others have made great progress in the last few years by understanding and harnessing the Transient Potential Receptor superfamily as regulators of cardiovascular function. Specifically, the investigators' laboratory has explored the role the vanilloid 2 (TRPV2) subtype plays in regulating calcium handling and contractility. This work has led researchers to understand that TRPV2 modulates contractility via increasing calcium cycling in myocytes on a beat-to-beat basis.

The investigators have used probenecid, a generic, globally available drug with an extremely safe profile that has been used for decades as a treatment for gout, as a TRPV2 agonist. The investigators' work with this drug has demonstrated it to be a potent inotrope without apoptotic, chronotropic or arrhythmogenic effects in cardiomyocytes in vitro as well as in vivo murine and porcine models. These findings have been taken to the bedside with a recently published small phase 2 study of 20 adult patients with HFrEF (the ReProsper HF pilot study) where the investigators demonstrated a mean improvement in left ventricular systolic and diastolic function with no adverse effects after only 1 week of treatment. The use of probenecid in HFrEF was also indirectly supported by a recent retrospective study of approximately 40,000 patients in the Medicare database that found treatment with probenecid (not specifically for heart disease) was associated with a 9% decreased risk of HF hospitalization. These studies strongly argue for the safety and potential efficacy of probenecid to improve systolic function and the need for a larger study, and of longer duration that also evaluates functional and health status outcomes in addition to systolic function.

The overall objective of this study is the treatment of outpatient Veterans with NYHA II-III heart failure with reduced ejection fraction (HFrEF) with probenecid to improve systolic and health function. Specifically, the investigators are proposing a three-site double-blinded, randomized, placebo-controlled, trial that will assess whether oral probenecid administered at 1 gr. orally twice per day for 180 days in patients with NYHA II-III HFrEF improves systolic function as measured via ejection fraction with echocardiography (aim 1); improves functional status as measured by exercise stress testing (aim 2); and improves self-report heart failure specific health status as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) and overall health status measured by EQ5D (aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Have documented heart failure as a treated inpatient or outpatient diagnosis in the medical record.
* Left ventricular ejection 40% within the past 12 months either by echocardiogram, cardiac MRI, cardiac CT, nuclear imaging or cardiac catheterization.

NYHA class II-III

* On stable GDMT for at least 2 weeks (including at least an EBM dose of betablocker and RAAS inhibition) consistent with the EPHESUS trial criteria [16] or having a documented allergy or adverse reaction to betablocker and/or RAAS inhibition.
* Age 18 years or older.

Exclusion Criteria:

* Acute coronary syndrome or cardiac revascularization within the past 3 months.
* End stage renal disease with renal replacement therapy or creatinine clearance less than 30 ml/min [17].
* Cardiac resynchronization therapy within the past 3 months.
* Constrictive pericarditis or restrictive cardiomyopathy on cardiac imaging study (echocardiogram cardiac MRI, cardiac CT) within the last 12 months.
* Ablation for cardiac arrhythmias within the past month.
* Peripartum cardiomyopathy diagnosed within past 6 months. If LVEF is still 40% after 6 months of diagnosis, they can be enrolled into the study.
* Uncorrected cyanotic congenital heart disease.
* Severe right sided valvular disease and/or greater than moderate degree of stenotic or regurgitant left valvular disease.
* Terminal illness with expected survival of less than 12 months.
* Women who are pregnant, breast feeding, or plan to become pregnant during the study. All women in childbearing age will undergo baseline and quarterly urine pregnancy tests to ensure absence of pregnancy since the cardiometabolic assessments will be different during pregnancy.
* Oral therapy with probenecid for any indication during the preceding 3 months.
* Hypersensitivity to probenecid based on prior exposure.
* Inability to provide informed consent or study procedures due to dementia, unstable psychiatric disease, or other cause (e.g. inability to do perform exercise testing).
* Acute gout attack within the previous 3 months.
* History of uric acid kidney stones within the last year. Patient will be removed from the study if they develop urate kidney stones.
* History of blood diseases in the past year: Aplastic anemia, Hemolytic anemia, Leukopenia, Neutropenia, Pancytopenia, Thrombocytopenia or leukemia.
* Creatinine clearance (eGFR) <30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cardiac function | 6 months
  The main primary outcome is echocardiogram-derived EF. The investigators will use Definity echo contrast if adequate endocardial border definition cannot be ascertained for EF calculation in apical 4 and apical 2 using volumetric tracing analysis and modified Simpson's. The echosonographers from all sites will follow the same standard study ECHO procedure to obtain the views

SECONDARY OUTCOMES:
Change from baseline in exercise tolerance via a symptom-limited exercise test on a cycle ergometer | 6 months
  The investigators will perform a maximal bicycle exercise stress test (BEST) on a cycle ergometer (Ergocard II, Esaote) with 25-W workload increments at 3-minute intervals. to adapt to patients with low functional capacity as previously described and with all the standard precautions. Results will be converted to Vo2 max using standard formula and compared to baseline
Change from baseline in The Kansas City Cardiomyopathy Questionnaire (KCCQ) and EQ5D | 6 months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23 item instrument validated in stable and decompensated HF patients with HFpEF and HFrEF. The questionnaire takes 4-6 minutes to complete and reflects disease-specific health status over the prior two weeks.
  Overall health status (EQ5D) (Appendix) is a well-known generic measure of health status. It has 5 questions that address five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety or depression) with five levels ranging from 'no problems' to 'extreme problems' each

CONTACTS AND LOCATIONS:
Overall Officials: Jack Rubinstein, MD, Principal Investigator — Cincinnati VA Medical Center, Cincinnati, OH
Locations (5):
- United States (5):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rubinstein J, Robbins N, Evans K, Foster G, Mcconeghy K, Onadeko T, Bunke J, Parent M, Luo X, Joseph J, Wu WC. Repurposing Probenecid for the Treatment of Heart Failure (Re-Prosper-HF): a study protocol for a randomized placebo-controlled clinical trial. Trials. 2022 Apr 7;23(1):266. doi: 10.1186/s13063-022-06214-y. PMID 35392963

DOCUMENTS (1):
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT04551222/ICF_000.pdf